CLINICAL TRIAL: NCT01817790
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multi-Center Study to Assess the Efficacy of Once-Daily Fluticasone Propionate Aqueous Nasal Spray 200mcg for 14 Days on Ocular Symptoms Associated With Seasonal Allergic Rhinitis
Brief Title: Assessment of Fluticasone Propionate on Ocular Allergy Symptoms
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: RH01619
Record Dates: First submitted 2013-03-21; First posted 2013-03-25 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2014-04-03 (Estimated); Status verified 2013-12

CONDITIONS: Allergic Rhinitis; Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic; Rhinitis, Allergic, Seasonal | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluticasone propionate nasal spray (Experimental): Fluticasone propionate nasal spray with strength per dose of 50 mcg/spray. Two sprays of study treatment per nostril to be administered in morning.
  Interventions: Drug: Fluticasone propionate
- Placebo nasal spray (Placebo Comparator): Two sprays of placebo per nostril to be administered in morning.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluticasone propionate — Nasal spray formulation (200 mcg/day)
  Other Names: Flonase
  Arms: Fluticasone propionate nasal spray
Drug: Placebo — Vehicle for Fluticasone propionate aqueous nasal spray
  Arms: Placebo nasal spray

SUMMARY:
This study is designed to investigate the efficacy of fluticasone propionate (FP) on ocular symptoms associated with allergic rhinitis (AR).

DETAILED DESCRIPTION:
While the current FP approved indication for GSK marketed formulation is limited to the treatment of nasal symptoms, several large well-controlled studies in which FP maintained adequate control of nasal symptoms when administered in a dose of 200 micrograms (mcg) once-daily (QD) also suggested improvement in ocular symptoms. This study will employ a randomized, double-blind, parallel group, multi-center design that compares FP and placebo nasal sprays in subjects with seasonal allergic rhinitis (SAR) to assess the effectiveness on ocular symptoms associated with AR.

ELIGIBILITY:
Inclusion Criteria:

1. Participants with good general health (in the opinion of the investigator) with no clinically significant and relevant abnormalities of medical history
2. Participants with diagnosis of seasonal allergic rhinitis

   1. A clinical history (written or verbal confirmation) of allergic rhinitis with the seasonal onset and offset of nasal and ocular allergy symptoms during each of the last 2 mountain cedar pollen allergy seasons.
   2. A positive skin test reaction to (at least) the relevant allergen, mountain cedar pollen, as determined by the skin pricks method performed within 12 months of Visit 1).
3. Participants with allergic rhinitis symptom of at least moderate severity for randomization:

   1. An iTOSS of ≥ 4 and an iNCSS of ≥2 on the morning of randomization (Visit 3/Baseline).
   2. An averaged (rTOSS) of ≥ 4, and an averaged rNCSS of ≥2 for three of the five days during the placebo lead in
4. Participant residing within a geographical environment where exposure to mountain cedar pollen is significant during the entire study period.
5. Participant demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent/assent and has received a signed and dated copy of the informed consent/assent form. Children, ages 12 to 17 will be required to sign an assent form as part of the informed consent process.

Exclusion Criteria:

1. Participants with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
2. Participants with nasal disorders like:

   1. injury or surgery to their nose that the investigator believes would interfere with participation in the study.
   2. previously diagnosed with a severe physical obstruction of the nose (e.g., deviated septum) that could affect the deposition of double-blind intranasal study drug.
   3. Rhinitis medicamentosa
3. Participants who have historical or current evidence of clinically significant uncontrolled disease like asthma, cardiac arrhythmias, hypertension, diabetes mellitus, ocular herpes, glaucoma, hepatic or renal disease, malignancy etc.
4. Presence of or symptoms of an active bacterial or viral infection.
5. Participants who have conjunctivitis caused by an infectious agent.
6. Participants with current, single eye or bilateral cataracts or participants who had cataract surgery within/less than 3 months

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 626 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- PPD Corporate Headquarters, Wilmington, North Carolina, United States

REFERENCES:
- [Derived] Ratner P, Van Bavel J, Mohar D, Jacobs RL, Hampel F, Howland W, Karwal R. Efficacy of daily intranasal fluticasone propionate on ocular symptoms associated with seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2015 Feb;114(2):141-7. doi: 10.1016/j.anai.2014.11.012. PMID 25624132
- See also: Related References DeWester 2003 — http://www.ncbi.nlm.nih.gov/pubmed/14619333

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 6 clinical sites in the US.
Pre-assignment Details: Of the 855 participants screened, 626 were randomized in the study. Of the 229 participants not randomized into the study, 151 did not meet the study criteria; 3 developed AEs; 10 were lost to follow-up; 4 violated protocol; 28 withdrew consent; and the remaining 33 were not randomized for other reasons.
Groups:
- Fluticasone Propionate Nasal Spray: Two sprays of Fluticasone propionate nasal spray (50 mcg/spray) per nostril to be administered in morning (Total dose 200 mcg).
Period: Overall Study
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Started | 314 | 312
Completed | 310 | 304
Not Completed | 4 | 8
Not completed — Adverse Event | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 2 | 1
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Other: Could not attend appointment | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray | Total
Number analyzed (Participants) | 314 | 312 | 626
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.4 (14.55) | 40.5 (16.36) | 40.5 (15.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 212 | 201 | 413
  Male | 102 | 111 | 213

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Reflective Total Ocular Symptom Score (rTOSS)
Description: The Reflective Total Ocular Symptom Score (rTOSS) is the sum of 3 individual participant-assessed symptom scores (eye itching/burning, eye tearing/watering, and eye redness), each evaluated using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe, for a possible score of 0-9. Subjects completed rTOSS in the evening (PM rTOSS; 12 hours post morning nasal spray use) and once in the morning (AM score: prior to nasal spray use). Daily (i.e. during one dosing interval) rTOSS is defined as the average of the PM rTOSS and the AM rTOSS of the next day prior to AM dosing. The mean change from baseline in (daily, AM, PM) TOSS was calculated as the subject's treatment period mean (over 14 days; from Day 0 PM to Day 14 AM) minus the baseline period (placebo run-in) mean.
Time Frame: Baseline to 14 days
Population: All subjects who were randomized into the study and received at least one dose of study product were included in the intent-to-treat (ITT) population. This analysis was conducted on ITT population.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 312
Score on a scale | -0.91 (1.625) | -0.63 (1.525)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in Daily rTOSS between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p = 0.0024, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; Treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.36, 95% CI 2-sided [-0.59 to -0.13]

2. Secondary Outcome: Mean Change From Baseline in AM rTOSS
Description: rTOSS is the sum of 3 individual participant-assessed symptom scores (eye itching/ burning, eye tearing/watering, and eye redness), each evaluated using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe, for a possible score of 0-9. For AM rToss, subjects completed rTOSS in the morning (AM score: prior to nasal spray use). The mean change from baseline in AM rTOSS was calculated as the subject's treatment period mean (over 14 days) minus the baseline period (placebo run-in) mean.
Time Frame: Baseline to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 312
Score on a scale | -0.96 (1.627) | -0.68 (1.573)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in AM rTOSS between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p = 0.0057, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; Treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.33, 95% CI 2-sided [-0.56 to -0.10]

3. Secondary Outcome: Mean Change From Baseline in PM rTOSS
Description: rTOSS is the sum of 3 individual participant-assessed symptom scores (eye itching/ burning, eye tearing/watering, and eye redness), each evaluated using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe, for a possible score of 0-9. For PM rTOSS, subjects completed rTOSS in the evening, 12 hours post morning nasal spray use. The mean change from baseline in PM rTOSS was calculated as the subject's treatment period mean (over 14 days) minus the baseline period (placebo run-in) mean.
Time Frame: Baseline to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 312
Score on a scale | -0.87 (1.735) | -0.60 (1.577)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in PM rTOSS between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p = 0.0009, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; Treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.41, 95% CI [-0.65 to -0.17]

4. Secondary Outcome: Mean Change From Baseline in Individual AM Reflective Ocular Symptom Scores for Eye Itching/Burning
Description: The AM Reflective Ocular Symptom Score was assessed individually for eye itching/burning using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe, for a possible score of 0-9. For evaluation, subjects completed the scoring in the morning, prior to nasal spray use. The mean change from baseline in AM Reflective Ocular Symptom Score (eye itching and burning) was calculated as the subject's treatment period mean (over 14 days) minus the baseline period (placebo run-in) mean.
Time Frame: Baseline to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 312
Score on a scale | -0.35 (0.581) | -0.28 (0.553)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in AM reflective symptom scores for Eye itching/burning between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p = 0.0117, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; Treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.10, 95% CI 2-sided [-0.19 to -0.02]

5. Secondary Outcome: Mean Change From Baseline in Individual PM Reflective Ocular Symptom Scores for Eye Itching/Burning
Description: The PM Reflective Ocular Symptom Score was assessed individually for eye itching/burning using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe, for a possible score of 0-9. For evaluation, subjects completed the scoring in the evening, 12 hours post morning nasal spray use. The mean change from baseline in PM Reflective Ocular Symptom Score (eye itching and burning) was calculated as the subject's treatment period mean (over 14 days) minus the baseline period (placebo run-in) mean.
Time Frame: Baseline to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 312
Score on a scale | -0.33 (0.626) | -0.24 (0.554)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in PM reflective symptom scores for Eye itching/burning between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p = 0.0005, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; Treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.15, 95% CI [-0.23 to -0.06]

6. Secondary Outcome: Mean Change From Baseline in Individual AM Reflective Ocular Symptom Scores for Eye Tearing/Watering
Description: The AM Reflective Ocular Symptom Score was assessed individually for eye tearing/watering using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe, for a possible score of 0-9. For evaluation, subjects completed the scoring in the morning, prior to nasal spray use. The mean change from baseline in AM Reflective Ocular Symptom Score (eye tearing/watering) was calculated as the subject's treatment period mean (over 14 days) minus the baseline period (placebo run-in) mean.
Time Frame: Baseline to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 312
Score on a scale | -0.35 (0.596) | -0.24 (0.589)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in AM reflective symptom scores for Eye Tearing/Watering between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p = 0.0023, ANCOVA — p-value was not adjusted for multiple comparisons; Least Square Mean Difference = -0.13, 95% CI [-0.22 to -0.06]

7. Secondary Outcome: Mean Change From Baseline in Individual PM Reflective Ocular Symptom Scores for Eye Tearing/Watering
Description: The PM Reflective Ocular Symptom Score was assessed individually for eye tearing/watering using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe, for a possible score of 0-9. For evaluation, subjects completed the scoring in the evening, 12 hours post morning nasal spray use. The mean change from baseline in PM Reflective Ocular Symptom Score (eye tearing/watering) was calculated as the subject's treatment period mean (over 14 days) minus the baseline period (placebo run-in) mean.
Time Frame: Baseline to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 312
Score on a scale | -0.32 (0.653) | -0.19 (0.586)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in PM reflective symptom scores for Eye Tearing/watering between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value was nor adjusted for multiple comparisons; Linear Fixed-effect Model; Treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.18, 95% CI [-0.26 to -0.09]

8. Secondary Outcome: Mean Change From Baseline in Individual AM Reflective Ocular Symptom Scores for Eye Redness
Description: The AM Reflective Ocular Symptom Score was assessed individually for eye redness using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe, for a possible score of 0-9. For evaluation, subjects completed the scoring in the morning, prior to nasal spray use. The mean change from baseline in AM Reflective Ocular Symptom Score (eye redness) was calculated as the subject's treatment period mean (over 14 days) minus the baseline period (placebo run-in) mean.
Time Frame: Baseline to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 312
Score on a scale | -0.26 (0.597) | -0.17 (0.613)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in AM reflective symptom scores for Eye Redness between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p = 0.0304, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; Treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.10, 95% CI [-0.18 to -0.01]

9. Secondary Outcome: Mean Change From Baseline in Individual PM Reflective Ocular Symptom Scores for Eye Redness
Description: The PM Reflective Ocular Symptom Score was assessed individually for eye redness using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe, for a possible score of 0-9. For evaluation, subjects completed the scoring in the evening, 12 hours post morning nasal spray use. The mean change from baseline in PM Reflective Ocular Symptom Score (eye redness) was calculated as the subject's treatment period mean (over 14 days) minus the baseline period (placebo run-in) mean.
Time Frame: Baseline to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 312
Score on a scale | -0.22 (0.628) | -0.17 (0.635)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in PM reflective symptom scores for Eye Redness between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p = 0.0361, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; Treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.10, 95% CI [-0.19 to -0.01]

10. Secondary Outcome: Mean Change From Baseline in AM Pre-dose Instantaneous Total Ocular Symptom Scores (iTOSS)
Description: Instantaneous total ocular symptom scores (iTOSS) assessments are self perceived evaluation of symptom severity immediately before the dose (how the subject feels at that point in time). iTOSS (possible score of 0-9) is the sum of 3 individual participant-assessed symptom scores for eye itching/burning, eye tearing/watering, and eye redness each evaluated using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe. Mean changes from baseline were calculated as treatment period iTOSS minus baseline iTOSS.
Time Frame: Baseline to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 312
Score on a scale | -0.80 (1.443) | -0.55 (1.531)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in AM iTOSS between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p = 0.0129, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.28, 95% CI 2-sided [-0.50 to -0.06]

11. Secondary Outcome: Mean Change From Baseline in Reflective Nasal Congestion Symptom Score (rNCSS)
Description: The rNCSS is a participant perceived evaluation of overall congestion symptom severity (evaluated using a scale of 0=None, 1=Mild, 2=Moderate, or 3=Severe) which was completed once in the evening (PM), and once in the morning (AM). rNCSS is defined as the average of the PM rNCSS and the AM rNCSS of the next day prior to AM dosing. The mean change from baseline in rNCSS (daily, AM, PM)was calculated as the subject's treatment period mean (over 14 days; from Day 0 PM to Day 14 AM) minus the baseline period (placebo run-in) mean.
Time Frame: Baseline to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 312
Score on a scale | -0.34 (0.547) | -0.20 (0.443)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in rNCSS between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p = 0.0002, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.14, 95% CI 2-sided [-0.22 to -0.07]

12. Secondary Outcome: End-of-treatment Assessment of Response to Therapy for Ocular Symptoms
Description: Overall response to therapy assessment was done using a 7-point categorical scale in which participants rated their response to therapy as follows: +3 = Significantly Improved; +2 = Moderately Improved; +1 = Mildly Improved; 0 = No Change; -1= Mildly Worse; -2 = Moderately Worse; -3 = Significantly Worse.
Time Frame: Day 14
Population: All subjects who were randomized into the study and received at least one dose of study product were included in the intent-to-treat (ITT) population. This analysis was conducted on ITT population. In this outcome measure, in Fluticasone propionate group 313/314 participants, and in the placebo group 309/312 participants provided responses.
Measure: Number; unit: Participants
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 313 | 309
Participants
  Significantly improved | 22 | 16
  Moderately Improved | 76 | 59
  Mildly Improved | 79 | 71
  No change | 81 | 97
  Mildly Worse | 21 | 20
  Moderatly Worse | 24 | 24
  Significantly Worse | 10 | 22
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the end of treatment assessment of response between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p = 0.0118, Cochran-Mantel-Haenszel — p-value was not adjusted for multiple comparisons; Using this test controlling for investigative site. The response variable lied on ordinal scale of measurement

13. Secondary Outcome: Mean Change in Objective Assessment of Conjunctival Redness
Description: Conjunctival redness was evaluated as a clinical sign of SAR by the investigator. Scoring of severity was rated according to a 4-point scale: 0 = normal; 1 = Slightly pink; 2 = Moderately pink, some dilation; 3 = Intense red vessels, dilated.
Time Frame: Baseline to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 312
Score on a scale | -0.20 (0.815) | -0.15 (0.736)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in objective assessment of conjunctival redness between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p = 0.8586, ANCOVA; Least Square Mean Difference = -0.01, 95% CI 2-sided [-0.12 to 0.10]

14. Secondary Outcome: Mean Changes From Baseline in Mini Rhinoconjunctivitis Quality of Life Questionnaire (MiniRQLQ) Scores
Description: MiniRQLQ is a 14-item, disease-specific instrument for assessing the impact of allergic rhinitis on activities of daily living and overall well-being. It measures five domains of functional impairment that are most important to subjects with SAR: practical problems, nasal symptoms, eye symptoms, activity limitations, and other symptoms. Participants scored their degree of impairment on a seven-point scale. (0 - 6). Mini RQLQ final score is the average of sub-scales, ranges from 0 (best possible outcome) to 6 (worst possible outcome).
Time Frame: Baseline to 14 days
Population: All subjects who were randomized into the study and received at least one dose of study product were included in the intent-to-treat (ITT) population. This analysis was conducted on ITT population. For analysis of nose symptoms, eye symptoms, and other symptoms, data of one participant each from the two groups are unavailable.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 311
Score on a scale | -0.98 (1.311) | -0.49 (1.091)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in MiniRQLQ scores between the Fluticasone nasal spray and the placebo nasal spray; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; Treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.47, 95% CI 2-sided [-0.65 to -0.29]

15. Secondary Outcome: Mean Changes From Baseline in Individual MiniRQLQ Scores: Domain - Activities
Description: MiniRQLQ is a 14-item, disease-specific instrument for assessing the impact of allergic rhinitis on activities of daily living and overall well-being. Activity limitations is one of the domains of Mini RQLQ scores. Participants scored their degree of impairment on a seven-point scale (0 = not troubled, 6 = extremely troubled).
Time Frame: Baseline to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 311
Score on a scale | -0.93 (1.384) | -0.39 (1.269)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in 'Activities' domain of MiniRQLQ scores between the Flutical sone nasal spray and placebo nasal spray; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; Treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.49, 95% CI 2-sided [-0.68 to -0.30]

16. Secondary Outcome: Mean Changes From Baseline in Individual MiniRQLQ Scores: Domain - Practical Problems
Description: MiniRQLQ is a 14-item, disease-specific instrument for assessing the impact of allergic rhinitis on activities of daily living and overall well-being. 'Practical Problems' is one of the domains of Mini RQLQ scores. Participants scored their degree of impairment on a seven-point scale (0 = not troubled, 6 = extremely troubled).
Time Frame: Baseline to 14 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 314 | 311
Score on a scale | -1.04 (1.476) | -0.57 (1.258)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in 'Practical Problems' domain of MiniRQLQ scores between the Flutical sone nasal spray and placebo nasal spray; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; Treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.44, 95% CI 2-sided [-0.64 to -0.24]

17. Secondary Outcome: Mean Changes From Baseline in Individual MiniRQLQ Scores: Domain - Nose Symptoms
Description: MiniRQLQ is a 14-item, disease-specific instrument for assessing the impact of allergic rhinitis on activities of daily living and overall well-being. "Nose Symptoms" is one of the domains of Mini RQLQ scores. Participants scored their degree of impairment on a seven-point scale (0 = not troubled, 6 = extremely troubled).
Time Frame: Baseline to 14 days
Population: All subjects who were randomized into the study and received at least one dose of study product were included in the intent-to-treat (ITT) population. This analysis was conducted on ITT population. For analysis of nose symptoms, data of one participant each from the two groups are unavailable.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 313 | 310
Score on a scale | -1.09 (1.456) | -0.50 (1.257)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in 'Nose Symptoms' domain of MiniRQLQ scores between the Flutical sone nasal spray and placebo nasal spray; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; Treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.53, 95% CI 2-sided [-0.73 to -0.33]

18. Secondary Outcome: Mean Changes From Baseline in Individual MiniRQLQ Scores: Domain - Eye Symptoms
Description: MiniRQLQ is a 14-item, disease-specific instrument for assessing the impact of allergic rhinitis on activities of daily living and overall well-being. "Eye Symptoms" is one of the domains of Mini RQLQ scores. Participants scored their degree of impairment on a seven-point scale (0 = not troubled, 6 = extremely troubled).
Time Frame: Baseline to 14 days
Population: All subjects who were randomized into the study and received at least one dose of study product were included in the intent-to-treat (ITT) population. This analysis was conducted on ITT population. For analysis of eye symptoms, data of one participant each from the two groups are unavailable.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 313 | 310
Score on a scale | -0.98 (1.512) | -0.55 (1.284)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in 'Eye Symptoms' domain of MiniRQLQ scores between the Flutical sone nasal spray and placebo nasal spray; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value was not adjusted for multiple comparisons; Linear Fixed-effect Model; Treatment and site as fixed factors and baseline score as covariate; Least Square Mean Difference = -0.44, 95% CI 2-sided [-0.65 to -0.23]

19. Secondary Outcome: Mean Changes From Baseline in Individual MiniRQLQ Scores: Domain - Other Symptoms
Description: MiniRQLQ is a 14-item, disease-specific instrument for assessing the impact of allergic rhinitis on activities of daily living and overall well-being. "Other Symptoms" is one of the domains of Mini RQLQ scores. Participants scored their degree of impairment on a seven-point scale (0 = not troubled, 6 = extremely troubled).
Time Frame: Baseline to 14 days
Population: All subjects who were randomized into the study and received at least one dose of study product were included in the intent-to-treat (ITT) population. This analysis was conducted on ITT population. For analysis of "other symptoms", data of one participant each from the two groups are unavailable.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Number analyzed (Participants) | 313 | 310
Score on a scale | -0.89 (1.607) | -0.48 (1.294)
Statistical Analysis 1: Comparison: Fluticasone Propionate Nasal Spray vs Placebo Nasal Spray; Null hypothesis was that no difference exists in the mean change from baseline in 'Other Symptoms' domain of MiniRQLQ scores between the Flutical sone nasal spray and placebo nasal spray; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-value was not adjusted for multiple comparisons; Least Square Mean Difference = -0.42, 95% CI 2-sided [-0.64 to -0.21]

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of study, an average of 3 weeks.
Arm/Group | Fluticasone Propionate Nasal Spray | Placebo Nasal Spray
Serious Adverse Events (participants affected / at risk) | 0/314 | 0/312
Other Adverse Events (participants affected / at risk) | 8/314 | 8/312
OTHER ADVERSE EVENTS (reported when occurring in more than 0.3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluticasone Propionate Nasal Spray (N=314) | Placebo Nasal Spray (N=312)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Thirst (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Gastrointestinal Viral (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.